CLINICAL TRIAL: NCT01084044
Title: Effects of Ulinastatin on Coagulation in High Risk Patients Undergoing Off Pump Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2009-0420
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Occlusive Disease
MeSH Terms: interventions — urinastatin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ulinastatin (Experimental)
  Interventions: Drug: ulinastatin, saline solution
- saline solution (Active Comparator)
  Interventions: Drug: ulinastatin, saline solution
- Sugar pill (Placebo Comparator)
  Interventions: Drug: ulinastatin, saline solution

INTERVENTIONS:
Drug: ulinastatin, saline solution — the ulinastatin group receiving ulinastatin (300,000 unit after anesthesia induction and another 300,000 unit during Y- graft anastomosis, n = 40), the control group receiving the same volume of saline solution(n = 40)

SUMMARY:
Ulinastatin reduce the amount of bleeding and fibrinolysis in high risk patients undergoing off-pump coronary bypass surgery (OPCAB).

ELIGIBILITY:
Inclusion Criteria:

* Eighty high risk patients undergoing OPCAB (High risk patients: Euro score ≥ 6 , acute coronary syndrome, preoperative CK-MB increased over 5 times than normal value and high sensitivity CRP ≥2.0)

Exclusion Criteria:

* The patients who receive additional operations, the patients who don't agree to participate in this trial, the patients who has a past hypersensitive experience on Ulinastatin

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
ulinastatin | 24 hours after surgery
  The purpose of this study was to evaluate whether ulinastatin significantly affect on coagulation and blood loss in high risk patients undergoing off-pump coronary bypass surgery (OPCAB). - thrombin-antithrombin complex (TAT), prothrombin fragment 1+2(F1,2), platelet factor-4 (PF-4) , hemoglobin, platelet count, white blood cell differential count, prothrombin time (PT), partial prothrombin time (aPTT), amount of blood loss, transfusion, urine output and intravenous fluid input

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea